CLINICAL TRIAL: NCT02312635
Title: Augmentation of Cognitive Training in Children With TBI With D-Cyloserine
Acronym: DCS
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Robert F. Asarnow, Ph.D, Della Martin Professor of Psychiatry, Professor of Psychology, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R21HD076418-01A1 (NIH)
Record Dates: First submitted 2014-02-06; First posted 2014-12-09 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Traumatic Brain Injury
Keywords: cognitive rehabilitation, traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cogmed + D-cycloserine (Experimental): Partifcipants will receive 6 weeks of cogmed working memory training M-F for 45 min each day. Participants in this arm will also take drug Monday, Wednesday, Friday throughout 6 weeks.
  Interventions: Drug: D-Cycloserine; Behavioral: Cogmed Working Memory Training
- Cogmed + Placebo (Placebo Comparator): Participants will receive 6 weeks of cogmed training M-F and also take a placebo pill Monday, Wednesday, Friday throughout 6 week period.
  Interventions: Behavioral: Cogmed Working Memory Training

INTERVENTIONS:
Drug: D-Cycloserine — Half of the participants will be randomly chosen to receive the medication D-cycloserine in addition to the working memory program, while the other group will receive an inactive pill (placebo).
  Other Names: Drug Trade Name--Seromycin, (D-cycloserine)
  Arms: Cogmed + D-cycloserine
Behavioral: Cogmed Working Memory Training — Both arms of the study will receive Cogmed working memory training for 6 weeks, M-F.

SUMMARY:
Traumatic Brain Injury (TBI) is the most common cause of death and long-term disability in children. Much of the long-term disability stems from neurocognitive impairments that are not greatly helped by current cognitive training and pharmacological treatments for TBI related cognitive impairments. This study tests the hypothesis that a drug, D-cycloserine (DCS), will significantly enhance the effect of cognitive training in correcting cognitive impairments in children with moderate/severe TBIs.

In order to do so, study subjects who fit inclusion criteria, including those with moderate to severe TBI who show persistent working memory weaknesses based on a screening, will be recruited. They will have three visits to UCLA. During the first visit, subjects will undergo an MRI protocol before and after taking a pill (drug or placebo, blinded). They will also participate in a number of paper and pencil cognitive tests. Then subjects will be enrolled in a 6 week computerized cognitive training program (CogMed). They will also be prescribed a drug/placebo pill (depending on which group they are randomized into), which they'll have to take at regular intervals during the 6 weeks. They will have weekly check in phone calls or visits by a coach trained in the program to make sure they are following the study protocol accurately, to have their questions answered, and for motivation. At the end of the training period, subjects will return to UCLA to again complete the MRI protocol and cognitive testing. After three months of enrollment, they will have a final visit to UCLA, including only cognitive testing. A total of 30 subjects will be entered into the study.

DETAILED DESCRIPTION:
Study Design/Procedure: The proposed study uses a double blind, parallel, placebo control design to test the hypotheses that augmentation of suppressed NMDA receptor function following pediatric msTBI with D-cycloserine (DCS) will increase neural activation, and when used in conjunction with cognitive training will enhance the effect of cognitive training on working memory (WM). Participants who show WM weaknesses within 12 to 24 months post-injury will be randomly assigned to one of two arms in the proposed study. Weakness in WM is operationally defined as a working memory index (WMI) standard score below 90 or evidence of at least a 10-point discrepancy between IQ and WMI. Given the purpose of the study (improving working memory), there is little utility in including children who do no demonstrate weaknesses in WM. Participants in both treatment arms will complete baseline evaluations on the WM and executive functioning (EF) tests that assess generalization, and parents will complete questionnaires that assess WM and attentional functioning. (Note: participants who completed their 12-month RAPBI visit within three months of enrollment in the current project will complete only novel measures). All participants will then receive their first Cogmed training session. During this first visit, participants will be also complete our MRI protocol immediately before and two hours after the first dose of DCS or placebo to measure the acute physiological response to DCS. Both groups will then complete six weeks of Cogmed training and in addition either DCS or placebo. Cogmed training will be completed in the home, with the parent/guardian supervising completion. During the six weeks of training, both you and your child will speak with a coach once a week, who will guide your child through the program and help to monitor his/her progress. Participants will travel to UCLA half-way through their training to consult with one of the medical personnel regarding the medication and to note any side effects. At the end of the sixth week, participants will be retested on our MRI protocol and non-trained measures of WM and EF. Parents will complete the questionnaires that assess WM and attention. Three months after the termination of treatment, participants will again return to UCLA to complete one session of Cogmed training and will be retested on the non-trained measures of WM and EF. Their parents will complete questionnaires to assess the maintenance of training.

Intercurrent events: Participants in the proposed project will be at least 12 months post-TBI. It is unlikely that new treatments will be initiated during the 4.5 months they are enrolled in the proposed project. Nevertheless we will monitor the medical and behavioral treatments outside of our study to ensure that they are not confounds.

Cogmed Training: Participants will perform the Cogmed WM training program via web-based software on a personal computer. If they do not have a personal computer, we will provide them with a laptop to borrow for the six weeks of training. Participants will train for 45 minutes per day, five days per week, for six weeks. Memory stimuli are presented in a computerized system in a total of eight visuospatial and verbal WM training exercises. Each training exercise consists of 15 trials. The exercises are in a video game format-with colorful graphics and crisp sound. In one spatial WM exercise the child remembers the sequence in which rows of lights turn on; in a verbal WM exercise the child recalls numbers in the reverse order in which they are given. The child uses a computer mouse to click the answers and earns points for performing well. The exercises train the child to attend to the screen and to visualize the location and remember the stimuli. For each of the eight WM training exercises difficulty is adjusted by changing the number of stimuli to be remembered. Training is performed close to the capacity of the individual by using an adaptive staircase method that adjusts difficulty on a trial-by-trial basis. At the end of each training day an Improvement index is calculated that measures improvement during the training period. The Improvement index is based on the person's results on three exercises.

On the first visit to UCLA, a coach will meet with the child and parent/guardian to teach them how to use the Cogmed program. The coach may encourage use a reward system to motivate and reinforce the child for training. The coach set up weekly times to contact the family. During these calls, the coach will review the child's progress, offer encouragement, and download performance data. The results of the improvement index will be shared with parents or adult participants, similar to how standardized paper and pencil neurocognitive test results are shared in clinical settings.

DCS treatment: DCS can have opposing effects at low dose vs. high dose. In mouse cerebellar tissue there is an inverted U-shaped dose-response relationship. At low DCS concentrations, agonist activity may reflect binding to NMDA receptor (NMDAR) subunits. In contrast, at higher DCS concentrations antagonist effects may become prominent. Consistent with the above research, in both animal models and clinical applications, isolated low dose DCS treatments appear to have significant advantages over chronic treatment at higher doses. In animal models, a single dose of DCS reversed cognitive impairment produced by hippocampal lesions, anticholinergic agents, and early social deprivation. In healthy animals, a single dose of DCS enhanced extinction of conditioned fear performance on maze tasks, and visual recognition memory. Mice treated with a single, low-dose of DCS 24 or 72 hours after TBI exhibited significantly more rapid and complete recovery of motor and memory function compared with untreated controls. Tachyphylaxis rapidly develops with repeated dosing of DCS. A single dose of DCS administered within 30 minutes of extinction training increases 24 hour retention of fear extinction approximately 3-fold, whereas this effect was completely attenuated by 5 doses of DCS administered over 10 days preceding the extinction training.

We will use isolated, low doses of DCS in the proposed project. When used to treat psychiatric symptoms or cognitive impairments in children the typical dose is 50-100mg. A meta-analysis of the effect of DCS augmentation of fear extinction and exposure therapy did not find significant dose related effects across studies but in the one clinical study that systematically investigated doses, there was some evidence of greater efficacy with a higher dose. In the proposed study participants will receive 100 mg of DCS. The same meta-analysis found that the best effects were evident when DCS was administered either immediately before or after exposure training compared to a four hour delay. Animal models and human studies suggest that DCS does not affect performance during training; instead, it selectively improves memory consolidation for new learning typically assessed 24 hour after training. The acute physiological effects of DCS on brain activation, however, can be observed two hours after DCS administration on fMRI.

In the proposed study children will take a pill (DCS or placebo) every other day immediately prior to Cogmed training. Over six weeks of Cogmed training they will train 18 days after taking a pill and 12 days without taking a pill. This intermittent, isolated dosing should minimize tachyphylaxis and reduce the possibility that Cogmed training results in state dependent learning.

Double Blind: The UCLA pharmacy will fabricate identically appearing capsules for 100 mg of DCS and placebo. Only the research pharmacist will know whether a child is receiving DCS or Placebo. The child and parent, the Cogmed coach, research psychologists, and the clinicians monitoring side effects will not know what drug the child is receiving. If there are clinically significant side effects, the blind will be broken.

Safety monitoring: Children in the DCS and placebo arms will be seen by Drs. Giza or Choe, who are pediatric neurologists, or their nurse practitioner three to four weeks after the initiation of treatment. In addition, the Cogmed coach will probe for side effects on each coaching call. Side effects will be assessed using a structured instrument and open-ended clinician inquiry. While there are scales for rating stimulant-related adverse events, we are not aware of a broadly accepted tool for glutamatergic agonists. Therefore, we will modify the Physical Symptom Checklist developed for the Research Units on Pediatric Psychopharmacology, which includes a range of potential adverse events.

Maximizing compliance/minimizing attrition: Weekly phone calls will be used to check on progress with Cogmed and assess motivation/compliance. As noted above, the coach may recommend use of a reward system to motivate and reinforce training. Any problems or issues will also be discussed during this call, with regards to both Cogmed and medication side effects. Participants will also meet with medical personnel during the third or fourth week of training to discuss possible side effects.

ELIGIBILITY:
Inclusion Criteria:

* non-penetrating msTBI (intake or post-resuscitation GCS score between 3 and 12)
* 11 to 18 years of age
* between 12 and 24 months post-injury
* working memory index (WMI) standard score below 90 or evidence of at least a 10 point discrepancy between estimated IQ and WMI
* normal visual acuity or vision corrected with contact lenses/eyeglasses
* English skills sufficient to understand instructions and be familiar with common words (the neuropsychological tests used in this study presume competence in English).

Exclusion Criteria:

* tumor or severe seizures
* motor deficits that prevent the subject from being examined in an MR scanner (e.g. spasms)
* history of psychosis,
* ADHD
* Tourette's Disorder
* learning disability
* mental retardation, autism or substance abuse. The latter conditions are associated with cognitive impairments that might overlap with those caused by TBI.
* participants with any metal implants that prevent them from safely undergoing an MRI scan are excluded.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-12; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Cogmed Working Memory Training Program | 6 weeks
  All participants will complete the Cogmed working memory training program for 6 weeks, M-F, for 45 minutes each day. Memory stimuli are presented in a computerized system in a total of 8 visuo-spatial and verbal working memory training exercises. Each training exercise consists of 15 trials. For each of the 8 working memory training exercises difficulty is adjusted by changing the number of stimuli to be remembered. Training is performed close to the capacity of the individual by using an adaptive staircase method that adjusts difficulty on a trial-by-trial basis. At the end of each training day an Improvement Index is calculated that measure improvement during the training period. The Improvement Index is based on the participant's results on 3 exercises.

SECONDARY OUTCOMES:
Wide Range Assessment of Memory & Learning-2 | Baseline
  All participants will be administered this test as a measurement of their working memory at baseline, 6weeks and 3months.
Wide Range Assessment of Memory & Learning-2 | 6 weeks
  All participants will be administered this test as a measurement of their working memory at baseline, 6weeks and 3months.
Wide Range Assessment of Memory & Learning-2 | 3 months
  All participants will be administered this test as a measurement of their working memory at baseline, 6weeks and 3months.

OTHER OUTCOMES:
Parent Reports | Baseline
  Parent measures will be administered to assess working memory and attention functioning.
Parent Reports | 6 weeks
  Parent measures will be administered to assess working memory and attention functioning.
Parent Reports | 3 months
  Parent measures will be administered to assess working memory and attention functioning.
Structural & Functional MRI | Baseline
  Structural & Functional Magnetic Resonance Imaging will be completed on participant to get baseline scans before participants begin intervention.
Structural & Functional MRI | 6 weeks
  Structural & Functional Magnetic Resonance Imaging will be completed on participant to get 6 week follow up scans to determine if there were any changes in brain after 6 week drug and working memory task interventions.
Structural & Functional MRI | 3 months
  Structural & Functional Magnetic Resonance Imaging will be completed on participant to get 6 week follow up scans to determine if there were any changes in brain after 3 months post interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Robert F Asarnow, Ph.D., Principal Investigator — University of California, Los Angeles; Christopher Giza, M.D., Principal Investigator — University of California, Los Angeles; Lisa Moran, Ph.D., Study Director — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States